CLINICAL TRIAL: NCT02162641
Title: R-SeNSAR Feasibility Study: The Role of Sentinel Node Biopsy in Patients With Anal Cancer
Brief Title: Study to Determine the Feasibility of Sentinel Node Biopsy in Patients With Anal Cancer
Acronym: R-SeNSAR
Status: Withdrawn | Type: Observational
Why Stopped: The study was terminated early as it failed to recruit.
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Emmie Taylor, Clinical Trials Project Manager, The Christie NHS Foundation Trust
Other Study IDs: 13_DOG03_261; CFTSp081 (Other: Sponsor)
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Squamous Cell Carcinoma of the Anus
MeSH Terms: conditions — Anus Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- SCC of the anus
  Interventions: Procedure: Sentinel lymph node biopsy

INTERVENTIONS:
Procedure: Sentinel lymph node biopsy

SUMMARY:
The purpose of this study is assess the technical and operational feasibility of a specialised biopsy technique, sentinel lymph node biopsy (SLNB), in patients with anal cancer.

DETAILED DESCRIPTION:
SLNB is based on the premise that lymphatic dissemination from a tumour occurs in a stepwise fashion, with initial involvement of a primary node, called the sentinel node, before dissemination to the remainder of the lymphatic chain. If the sentinel node is histologically negative, then the remainder of the nodes in the same anatomic region will be at a lower (assumed to be minimal) risk of containing metastases. SLNB is part of standard care for patients with malignant melanoma and with breast cancer but has yet to be prospectively evaluated in patients with anal cancer.

Currently, the standard way to treat patients with anal cancer is to deliver a combination of chemotherapy and radiation to the tumour at the anus together with 'preventative' (prophylactic) radiotherapy to the lymph glands of the groin and pelvis. There is a growing perception for the need to reduce the morbidity of radiotherapy i.e. current regimens over-treat the patient and one approach is to reduce radiotherapy volume and/or dose where there is an absence or very low risk of nodal metastases.

This feasibility study is a vital first step in informing the design of a larger study examining the role of SLNB in clinical decision-making and outcomes for patients with anal cancer. In this trial eligible patients will attend for lymphoscintigraphy, to locate the lymph node, before sentinel lymph node removal by surgery. Detection rate of the sentinel node(s) will be the key outcome for the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with squamous cell carcinoma (SCC) of the anus (any T size and/or those with recurrent disease)
* Equivocal lymph node involvement on standard CT staging or magnetic resonance (MR) staging or PET-CT scan, as determined by the anal cancer multidisciplinary team (MDT)
* Age >= 18 years
* Written informed consent provided by the patient

Exclusion Criteria:

* Patients with unequivocal lymph node involvement on standard CT staging or MR staging, as determined by the anal cancer MDT.
* Unfit for surgical biopsy
* Patients undergoing palliative treatment
* Previous pelvic or inguinal area radiotherapy
* Other coincident cancers
* Previous inguinal surgery (e.g. hernia repair) with mesh insertion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with squamous cell carcinoma (SCC) of the anus with clinically negative or equivocal nodal involvement; and for consideration of chemo-radiotherapy, local excision or salvage surgery treatment. The majority will be initial presentations, but patients with recurrent disease may also be considered.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The proportion of nodes detected will be expressed per inguinal nodal basin and per number of patients | Day 0 (Day of SLNB)

SECONDARY OUTCOMES:
Micro-metastatic disease within sentinel nodes | Days 7 to 10
Surgical complications | Up to 15 weeks after SLNB
  To include wound healing assessment and assessment of pain
Delays in receiving radiotherapy treatment | 15 weeks after SLNB
  Any delay greater than 37 days from presentation to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Renehan, Study Chair — The Christie NHS Foundation Trust